CLINICAL TRIAL: NCT00269555
Title: Effects of a Genistein Combined Polysaccharide (GCP) on Patients With a Diagnosis of Prostate Cancer on Active Surveillance.
Brief Title: Effects of GCP on Prostate Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Dr. Robert Hackman, University of California, Davis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200412146
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Prostate Specific Antigen; C04.588.945.440.770
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — genistein combined polysaccharide

INTERVENTIONS:
Drug: Genistein Combined Polysaccharide (GCP)

SUMMARY:
Genistein Combined Polysaccharide (GCP) is derived from adding soy powder to shiitake mushrooms. This concentrated mixture is currently being sold in Japan and the United States and is thought to possibly contain properties that may be useful in treating certain types of cancer.

ELIGIBILITY:
Inclusion Criteria:

Participants must be male and have a pathological diagnosis of prostate cancer.

No treatment (surgery [RRP], radiation, or hormones) prior to study entry.

The patient has decided, after consultation with his own doctor, to have no treatment intervention (surgery [RRP], radiation, or hormones) for the next six months.

PSA between 2.0 and 10.0 ng/ml.

If PSA is >10.0, patient must have been on Active Surveillance for 12 months prior to study initiation.

No known allergy to soy or soy products.

The patient is not currently taking more than 2 grams of genistein a day in nutritional or diet enhancing supplements (OTC supplements).

-

Exclusion Criteria:

No pathological documentation of prostate cancer.

Allergy to soy or soy products

Prior history of treatment for prostate cancer.

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62
Dates: Start 2004-05; Primary Completion 2006-01 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Reduction in PSA serum levels.

SECONDARY OUTCOMES:
Stabilization of PSA serum levels.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hackman, PhD, Principal Investigator — University of California, Davis; Ralph W deVere White, MD, Study Director — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

REFERENCES:
- [Background] deVere White RW, Hackman RM, Soares SE, Beckett LA, Li Y, Sun B. Effects of a genistein-rich extract on PSA levels in men with a history of prostate cancer. Urology. 2004 Feb;63(2):259-63. doi: 10.1016/j.urology.2003.09.061. PMID 14972467